CLINICAL TRIAL: NCT03697005
Title: One Year Clinical Evaluation of Pressed BioHPP Polyether Ether Ketone (PEEK)-Based Versus Zirconia-Based Single Crowns (Randomized Controlled Clinical Trial)
Brief Title: One Year Clinical Evaluation of Pressed BioHPP Polyether Ether Ketone (PEEK)-Based Versus Zirconia-Based Single Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Ezzat Mohamed Ali El-shimy, Assistant lecturer, fixed prosthodontic department, faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-40
Record Dates: First submitted 2018-09-28; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Clinical Performance; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Composite Resins; Dental Porcelain

STUDY DESIGN:
Intervention Model Description: patients requiring posterior single crowns.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinding (trial participants and outcome assessor)
  * Dental colleague assessors who are blinded about the aim of the study and participant's allocation will be responsible for assessing the outcomes of this study.
  * The level of intra- and inter-examiner reliability will be determined for each assessor by the performance of a calibration session prior to the start of the trial. A training exercise to the assessors with the main investigator will help to standardize measurement techniques and parameters. An interactive calibration session will enable the investigator to quantitate the measurement variability among and between assessors and enable the optimization of the measurement process. The main supervisor will solve any conflict that may arise between the assessors by repeating the assessing and giving the final opinion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioHPP PEEK single posterior crowns (Experimental): BioHPP PEEK copings veneered with composite resin
  Interventions: Other: BioHPP PEEK single posterior crowns
- zirconia-based single posterior crowns (Active Comparator): yttria stabilized tetragonal zirconia used as copings to be veneered with porcelain
  Interventions: Other: zirconia-based single posterior crowns

INTERVENTIONS:
Other: BioHPP PEEK single posterior crowns — BioHPP is a 20% ceramic reinforced, semicrystalline, thermoplastic and radiolucent polymeric material, used for fabrication of high strength fixed and removable prostheses. it has advantages of bio-compatibility, low density, light weight, shock absorption.
  Other Names: BioHPP PEEk copings veneered with composite resin
  Arms: BioHPP PEEK single posterior crowns
Other: zirconia-based single posterior crowns — ZrO2, a ceramic material used for medical devices, displays good esthetic appearance, high mechanical strength, and high biocompatibility and is used in a wide range of indications, such as frameworks, implants, and abutments. In addition, it's very good long-term stability and reliability was proven in a 10-year clinical study. These excellent material properties and the transformation behavior are explained by the yttrium oxide stabilization of ZrO2.
  Other Names: zirconia copings veneered with porcelain
  Arms: zirconia-based single posterior crowns

SUMMARY:
The clinical performance (using the modified Ryge criteria) and patient satisfaction ( using VAS questionnaire) of pressed BioHPP PEEK based posterior single crowns compared to zirconia based crowns are questionable as the peek is considered as a new material and need to be tested for future clinical application.

DETAILED DESCRIPTION:
The study is held to evaluate the clinical performance (using the modified Ryge criteria) and patient satisfaction ( using VAS questionnaire) of pressed BioHPP PEEK based posterior single crowns compared to zirconia based crowns after one year follow-up. Patients requiring posterior single crowns are collected. After teeth preparation to receive single full coverage crowns, secondary impressions were taken. The patients were divided randomly into two groups ;one group will receive pressed BioHPP PEEK single crowns (the intervention) and the other group will receive veneered zirconia single crowns (the control). Fracture of restorations (1ry outcome) using modified Ryge criteria and the marginal adaptation (2ry outcome) using modified Ryge criteria and finally the patient satisfaction (3ry outcome) using a questionnaire, all outcomes will be evaluated every 2 months with total period of follow-up of one year.

ELIGIBILITY:
Inclusion Criteria:

1. From 18-50 years old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations
3. Psychologically and physically able to withstand conventional dental procedures
4. Patients with teeth problems indicated for single posterior crowns:

   1. Badly decayed teeth
   2. Teeth restored with large filling restorations
   3. Endodontically treated teeth
   4. Malformed teeth
   5. Malposed teeth (Tilted, over-erupted, rotated, etc.)
   6. Spacing between posterior teeth
5. Able to return for follow-up examinations and evaluation

Exclusion Criteria:

1. Patient less than 18 or more than 50 years
2. Patient with active resistant periodontal diseases
3. Patients with poor oral hygiene and uncooperative patients
4. Pregnant women
5. Patients in the growth stage with partially erupted teeth
6. Psychiatric problems or unrealistic expectations
7. Lack of opposing dentition in the area of interest
8. Failed endodotically treated teeth; short or overextended, narrow, missed canal, ledge or perforated teeth (even if no clear symptoms for failure)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Fracture | one year
  Fracture of the single crowns assessed by modified Ryge criteria (Alpha, Bravo, Charlie and Delta)

SECONDARY OUTCOMES:
Marginal adaptation | one year
  Marginal adaptation assessed by modified Ryge criteria (Alpha, Bravo, Charlie and Delt

OTHER OUTCOMES:
patient satisfaction | one year
  patient satisfaction assessed by VAS questionnaire

IPD SHARING:
Plan to Share IPD: No